CLINICAL TRIAL: NCT02759406
Title: Evaluation of the Palmaz Mach-5 Grooved Bare Metal Coronary Stent System Versus the Palmaz Bare Metal Coronary Stent System in Patients With Symptomatic Ischemic Heart Disease: A Safety and Performance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palmaz Scientific (Industry)
Collaborators: ClinLogix. LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mach-5
Record Dates: First submitted 2016-04-27; First posted 2016-05-03 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

ARMS (2):
- Mach-5 Grooved (Experimental): grooved
  Interventions: Device: coronary stent
- Mach 5 Bare Metal (Experimental): bare metal
  Interventions: Device: coronary stent

INTERVENTIONS:
Device: coronary stent

SUMMARY:
This is a six (6) month, randomized, un-blinded, study to assess the safety and performance of the Palmaz Mach-5 Grooved Coronary Stent System vs. the Palmaz Bare Metal Coronary Stent System.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients of any race greater than or equal to 18 years and of legal consent
2. Patients must be willing to comply with the specified follow-up evaluation schedule
3. Patients who sign an informed consent (signed and dated) prior to any study-related evaluation or procedure.
4. Patients who are willing to undergo a follow-up coronary angiogram and Endovascular Imaging via Optical Coherence Tomography
5. Patients willing to be maintained on Aspirin and Clopidogrel bisulfate (Plavix) for ninety (90) days post procedure.
6. Patients with a de novo coronary lesion causing angina and/or a positive function test
7. Patients who are eligible for percutaneous coronary interventions
8. Low risk NSTEMI defined as patients with ACS, unstable angina, positive cardiac biomarkers and hemodynamically stable as assessed by the Investigator.
9. Patients with an acceptable risk for coronary bypass graft surgery (CABG)

Intra-Procedure Angiographic Criteria:

1. Single de novo target lesion >50% diameter stenosis by angiography
2. Single target vessel 2.75 to 3.25 mm diameter
3. Lesion length of 14 to 20mm which is suitable for Palmaz Mach-5 Grooved Coronary Stent System or the Palmaz Bare Metal Coronary Stent System.

Exclusion Criteria:

1. Known allergy or sensitivity to cobalt chromium (CoCr) alloy or its components.
2. Known sensitivity or allergy to aspirin, radiographic contract agents (that cannot be pre-treated adequately).
3. Patients unable to tolerate anticoagulant therapy or antiplatelet therapy.
4. History of bleeding or known coagulopathy.
5. Patients with thrombocytopenia and or neutropenia.
6. More than one stenosis >50% in target vessel.
7. Lesion in aortic ostium.
8. Left main or LAD, CX lesions within 2-mm from the origin.
9. Ejection Fraction <45%.
10. STEMI in evolution.
11. Disabling stroke within previous 30 days.
12. Patients currently enrolled in another Investigational device or drug study.
13. Previous enrollment in this study.
14. Women who are currently pregnant. (A negative pregnancy test for female subjects of child bearing potential is required within 24 hours of procedure.)
15. Known or suspected active systemic infection.
16. Evidence of severe or uncontrolled systemic diseases, including chronic renal insufficiency, or any condition which in the Investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-09; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
late lumen loss rate by Quantative/ Qualtative Cornary Angiographia | 6 month
total percentage of strut coverage by Optical Coherence Tomography analysis | 6 month
Primary safety endpoint is the occurrence of adverse events associated with the Investigational and comparator devices. | 6 month
binary restenosis rate by Quantative/ Qualtative Cornary Angiographia | 6 month